CLINICAL TRIAL: NCT02867696
Title: Effect of a Technology-Based Intervention on Weight Change Post-Bariatric Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO14060446
Record Dates: First submitted 2016-05-05; First posted 2016-08-16 (Estimated); Last update posted 2021-08-10 (Actual); Status verified 2020-03

CONDITIONS: Motor Activity; Weight Loss
Keywords: Bariatric Surgery; Physical Activity; Weight Management; Weight Loss
MeSH Terms: conditions — Motor Activity; Weight Loss | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Care (Active Comparator): Standard Care serves as the no treatment control in this project. Participants in this group will receive the typical care from their surgeon following bariatric surgery. No additional interventions will be given to participants randomized to this group.
  Interventions: Other: Standard Care
- Technology-based Intervention (TECH) (Experimental): TECH is the experimental group in this project. A minimal-contact technology-based intervention for weight management will be given to this group in addition to the standard or typical care received from their surgeon following bariatric surgery.
  Interventions: Behavioral: Technology-based Intervention (TECH)

INTERVENTIONS:
Other: Standard Care — Subjects in this arm will receive the standard care that is provided by their bariatric surgical team following bariatric surgery.
  Arms: Standard Care
Behavioral: Technology-based Intervention (TECH) — Dietary recommendations: based on the subjects' baseline body weight, with calorie goals ranging from 1200-2100 kcal/day.
  The physical activity component: unsupervised home-based exercise program. Intensity/Mode: aerobic physical activity recommended at a moderate intensity. Prescription: progress to 250 min/wk by 13th week of the intervention.
  Self-monitoring: Jawbone UP3 System includes a wearable device to monitor physical activity and energy expenditure that will transmit real-time feedback on calories expended and physical activity directly to a smart phone. An integrated digital smart scale will also be provided.
  Contact: scheduled intervention telephone call: Month 1: One call per week for the first 4 weeks of the study; Months 2-6: One call per month.
  Arms: Technology-based Intervention (TECH)

SUMMARY:
The primary aim of this study is to examine the effect of applying a minimal contact technology-based intervention (TECH) at 1-year post-bariatric surgery on weight change compared to Standard Care. Forty participants at 1-year post bariatric surgery will be randomized to TECH or Standard Care for a period of 6 months (12 to 18 months post-surgery). Analyses will be conducted to compare these interventions for differences in body weight, body composition, fitness, physical activity, engagement, psychosocial measures, and intervention cost and cost-effectiveness of each approach. TECH will consist of a wearable monitor that provides feedback on energy expenditure and physical activity, electronic tracking of dietary intake, and integration of an electronic scale to provide comprehensive feedback to the participant on all components of weight management. TECH participants will receive a monthly telephone call from the intervention staff to provide guidance on their weight management efforts.

DETAILED DESCRIPTION:
This randomized controlled trial will examine the effect of a minimal contact technology-based system in comparison to standard care on body weight in adults 1 year post-bariatric surgery. This 6 month intervention will be conducted at the University of Pittsburgh, Physical Activity and Weight Management Research Center. Eligible participants who obtain physician's consent will undergo baseline assessments. Assessments will be described in further detail below.

Eligible participants who complete all baseline assessment procedures will be randomized to one of two intervention groups: The minimal contact technology-based intervention using the Jawbone UP3 System combined with a monthly intervention telephone call (TECH), or Standard Care.

Standard Care serves as the no treatment control in this project. Participants in this group will receive the typical care from their surgeon following bariatric surgery. No additional interventions will be given to participants randomized to this group.

TECH Intervention: TECH is the experimental group in this project. A minimal-contact technology-based intervention for weight management will be given to this group in addition to the standard or typical care received from their surgeon following bariatric surgery. The following information outlines the protocol for this intervention group.

Dietary Component: Dietary recommendations will be based on the subjects' baseline body weight, with calorie and fat intake goals ranging from 1200-2100 kcal/day and 20-30% of daily calories respectively. The calorie goals are based on intake recommendations that have been shown to result in successful short-term weight loss with fat intake goals consistent with the USDA Dietary Guidelines. To facilitate adoption and maintenance of these dietary intake goals, participants will be provided with meal plans and sample recipes. In addition, participants will be taught how to read food labels and will be provided with The Calorie King Calorie, Fat, and Carbohydrate Counter to facilitate self-monitoring of calorie and fat intake. Intervention lessons will be sent to the participants via email and will also include information related to behavior strategies for achieving the desired calorie and fat intake goals.

Physical Activity Component: The physical activity component will include an unsupervised home-based exercise program. Participants will be asked to perform aerobic physical activity recommended at a moderate intensity defined as 3-6 metabolic equivalents (METS). This intensity is similar to brisk walking, however can be achieved through aerobic-based activities of the participants' choice. Equipment will not be provided to the participants. To facilitate adoption of this intensity of physical activity, participants will be provided both a target heart rate (60-70% of age-predicted maximal heart rate) and rating of perceived exertion (11-13 on the 15-category Borg Scale). Baseline physical activity participation will be evaluated and intervention recommendations will be prescribed to progress to 250 minutes per week by 13th week of the intervention, which is consistent with the recommendations of the American College of Sports Medicine (ACSM). Participants will be encouraged to complete the prescribed doses of physical activity each week, with daily goals achieved by performing the activity in one continuous bout or accumulated across several shorts bouts that are each at least 10 minutes in duration. Intervention lessons will be sent to the participants via email and will also include information related to behavior strategies for achieving the desired activity goals for this study.

Participants in this group will be provided with the Jawbone UP3 System. The Jawbone UP3 System includes a wearable device to monitor physical activity and energy expenditure that will transmit real-time feedback on calories expended and physical activity directly to a smart phone containing the web-interface/application. In addition, the smart phone supports self-monitoring of dietary behaviors and body weight to provide real-time feedback of goal achievement. A digital smart scale will also be provided to TECH participants. The smart scale (Withings®, Inc.) transmits objective measures of body weight directly to a smart phone application which also interfaces with the Jawbone UP3 System. All technology tools (UP3 system in combination with the smart scale) will allow for self-monitoring of energy expenditure, energy balance, physical activity, dietary intake, and body weight to occur in real-time and within an integrated system. Participants will attend one introductory session in which a tutorial of the components of the Jawbone UP3 System and smart scale will be provided. Individuals will be given confidential login codes which will provide access to the websites and smart phone applications. Login procedures as well as uploading data and Bluetooth® syncing of the technology components will be demonstrated. Detailed written instructions will also be given illustrating these procedures. Additionally, a follow-up call within 1 week of the initial meeting will occur to make sure that all technology components are working properly.

TECH will also initially receive a one-hour lesson on basic guidelines of the weight management intervention. At this time, caloric goals and weekly physical activity recommendations will be explained. To support weight loss behaviors, participants will be encouraged to use the Jawbone UP3 System and smart scale to self-monitor dietary intake, physical activity, and body weight.

Participants in TECH will also receive a scheduled intervention telephone call from a study coach on the following schedule:

-Month 1: One call per week for the first 4 weeks of the study. This will support the participants with making changes to their lifestyle behaviors as a part of the intervention. Additionally, this call will be used to ensure that the technology is functioning properly and that it is being used as intended by the study.

Months 2-6: One call per month. This call will be used to provide continued intervention support in addition.

These telephone calls will take approximately 10-15 minutes and will be completed by a member of the intervention staff that is experienced using the Jawbone UP3 System and smart scale and is trained in delivering behavioral telephone interventions. Strategies to overcome weight-loss barriers will be primarily discussed, and a standardized script will serve as a guide to address technical difficulties using the UP3 System and smart scale, frequency of technology usage, participant goals, barriers to diet and physical activity, and monitoring of body weight. Interventionists will have access to the information uploaded to the web-interfaces from the UP3 System and smart scale, and this will allow the interventionist to review this information prior to facilitating interactions with participants during the telephone calls. The length of each telephone intervention will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-60 years.
* 1-year post-bariatric surgery.
* Able to walk at 3 miles per hour during a cardiorespiratory fitness test.

Exclusion Criteria:

* Reports not having access to a computer, access to the Internet, email, or the availability to download software onto a computer.
* Reports not having a smart phone device that is compatible with the Jawbone UP3 System that will be examined in this study.
* Has a physical limitation that would prevent engaging in physical activity.
* Reports being treated for a current medical condition that could affect body weigh (diabetes mellitus, cancer, chronic renal insufficiency, hyperthyroidism, hypothyroidism, chronic liver disease).
* Reports current congestive failure, angina, uncontrolled arrhythmia, symptoms indicative of increased risk of an acute cardiovascular event, coronary artery bypass grafting or angioplasty, prior myocardial infarction, and conditions requiring anticoagulation therapy (deep vein thrombosis).
* Has a resting systolic blood pressure ≥ 150 mmHg or resting diastolic blood pressure of ≥100 mmHg or taking medication to control blood pressure that affects heart rate.
* Reports being treated for a psychological issue (i.e., depression, bipolar disorder, etc).
* Taking prescription or over-the-counter medications that affect body weight and metabolism.
* Currently participating in an exercise or weight control study or a current participant in a commercial weight reduction program.
* Currently being treated for an eating disorder.
* Currently pregnant, pregnant in the last 6 months, breast feeding in the last 3 months, lactating, to planning on becoming pregnant in the next 6 months.
* Planning on relocating outside of the greater Pittsburgh area within the next 6 months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-01; Primary Completion 2021-04-29 (Actual); Study Completion 2021-04-29 (Actual)

PRIMARY OUTCOMES:
To examine the effect of applying a minimal contact technology-based intervention (TECH) at 1-year post-bariatric surgery on weight change compared to Standard Care over the subsequent 6 months. | 1 year after bariatric surgery - months 12-18 (6 month intervention period)
  Body Weight (5 minutes; 0, 3, 6 months): Body weight will be measured to the nearest 0.1 kg on a Tanita WB-110A digital scale (Tanita Corporation; Arlington Heights, IL). Measures will be taken in a light-weight hospital gown with shoes and accessories removed.

SECONDARY OUTCOMES:
To examine the effect of TECH and Standard Care on change in body composition. | 1 year after bariatric surgery - months 12-18 (6 month intervention period)
  Regional Adiposity by Anthropometry (5 minutes; 0, 6 months): Taken in a lightweight hospital gown and measured to the nearest 0.1 cm using a Gulick tape measure. Waist circumference will be taken from the front at the level of the iliac crest. Hip circumferences will be taken from the side while making a horizontal circumference at the maximal protrusion of the gluteal muscles.
  Body Composition (30 minutes total; 0, 6 months): Body composition will be assesses using 2 methods (1) bioelectrical impedance analysis (BIA), and (2) dual xray absorptiometry (DXA).
To examine the effect of TECH and Standard Care on change in cardiorespiratory fitness. | 1 year after bariatric surgery - months 12-18 (6 month intervention period)
  Cardiorespiratory Fitness: (40 minutes; 0, 6 months): Subjects will complete a graded exercise test on a treadmill using indirect calorimetry to measure peak oxygen consumption. With peak oxygen used to define cardiorespiratory fitness.
To examine the effect of TECH and Standard Care on change in physical activity (Paffenbarger) | 1 year after bariatric surgery - months 12-18 (6 month intervention period)
  Physical activity (0, 3, 6 months) will be assessed using self-report questionnaire: Paffenbarger Physical Activity Questionnaire (Paffenbarger 1986)
  This questionnaire will provide minute/week data on moderate-to-vigorous physical activity performed with walking, stair climbing, and other recreational/fitness activities.
To examine the effect of TECH and Standard Care on change in physical activity (GPAQ) | 1 year after bariatric surgery - months 12-18 (6 month intervention period)
  Physical activity (0, 3, 6 months) will be assessed using self-report questionnaire: Global Physical Activity Questionnaire (GPAQ)
  This questionnaire will provide minute/week data on occupational, household, leisure and recreational, and transportation physical activities.
To examine the effect of TECH and Standard Care on change in physical activity (objective monitor) | 1 year after bariatric surgery - months 12-18 (6 month intervention period)
  Physical activity (0, 3, 6 months) will be assessed using an objective physical activity monitor: Sensewear Pro Armband
  This monitor (worn for 7 consecutive days) will provide minute/week data on sedentary, light, and moderate-to-vigorous physical activity.
To examine the effect of TECH and Standard Care on change in sedentary behavior. | 1 year after bariatric surgery - months 12-18 (6 month intervention period)
  Sedentary Behavior (0, 3, 6 months) will be assessed using self-report questionnaire: Sedentary Behavior Questionnaire
  This questionnaire will provide data on total time spent in sedentary activities on week and weekend days.
To examine the effect of TECH and Standard Care on change in dietary intake. | 1 year after bariatric surgery - months 12-18 (6 month intervention period)
  The Block Food Frequency Questionnaire will be used to assess the usual frequency of specific foods and typical portion sizes.
To examine the effect of TECH and Standard Care on change in eating behavior. | 1 year after bariatric surgery - months 12-18 (6 month intervention period)
  The Eating Behavior Inventory will be used to assess eating behaviors and behaviors that may be related to successful weight loss such as self-monitoring of intake, refusing food, shopping practices, and emotional eating.
To examine the effect of TECH and Standard Care on change in exercise barriers. | 1 year after bariatric surgery - months 12-18 (6 month intervention period)
  The Exercise Outcome, Expectations and Barriers questionnaire will be used to assess physical activity and exercise engagement and barriers.
To examine the effect of TECH and Standard Care on change in physical activity self-efficacy. | 1 year after bariatric surgery - months 12-18 (6 month intervention period)
  The Physical Activity Self-Efficacy questionnaire will be used to assess the subjects' confidence and self-efficacy for being physically active.
To examine the effect of TECH and Standard Care on change in health perception. | 1 year after bariatric surgery - months 12-18 (6 month intervention period)
  The SF-36 questionnaire will be used to assess perceptions of their health.
To examine the effect of TECH and Standard Care on change in weight loss and diet expectations and barriers | 1 year after bariatric surgery - months 12-18 (6 month intervention period)
  The Weight Loss Expectations and Barriers questionnaire will be used to assess perceptions around benefits and difficulties of weight loss and weight management.
To examine the effect of TECH and Standard Care on change in cognitive restraint and disinhibition with eating behaviors | 1 year after bariatric surgery - months 12-18 (6 month intervention period)
  The 3-Factor Eating/Eating Inventory questionnaire will be used to assess cognitive restraint, disinhibition, and perceived hunger related to eating behaviors.
To examine the effect of TECH and Standard Care on change in body image | 1 year after bariatric surgery - months 12-18 (6 month intervention period)
  The Multidimensional Body-Self Relations/Body Image Scale questionnaire will be used to assess body image.
To examine the effect of TECH and Standard Care on change in depression symptoms | 1 year after bariatric surgery - months 12-18 (6 month intervention period)
  The CES-D (short form) will be uses to assess depressive symptoms.
To examine satisfaction related to technology usage for weight management | 1 year after bariatric surgery - months 12-18 (6 month intervention period) - collected at 6 months
  A survey will be administered to determine subject satisfaction related to technology usage during the study and interest in potential continued usage. This will be administered at 6 months to the TECH group only.
To conduct analyses to examine the cost and cost effectiveness of TECH and Standard Care interventions. | 1 year after bariatric surgery - months 12-18 (6 month intervention period)
  Analyses of cost will be broken down by payer, participant, and societal perspectives.
  Payer costs referring to labor (time, wage) plus non-labor (materials, fixed costs, intervention-specific materials) costs.
  Participant costs including Time in minutes (in-person, phone calls), Attendance (transit minutes, inperson attendance), Wage based on BLS average, and Transport (transportation costs).
  Total Social costs will be the sum of Payer and Participant costs.

CONTACTS AND LOCATIONS:
Overall Officials: Renee J. Rogers, Ph.D., Principal Investigator — University of Pittsburgh
Locations (1):
- Physical Activity and Weight Management Research Center / University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
It is not known at this time if data will be shared at the conclusion of the project.